CLINICAL TRIAL: NCT03155971
Title: Efficacy and Safety of Paclitaxel-Coated Balloon Catheter in Patients With Long De Novo Lesions of Main Coronary Arteries
Brief Title: PCB for Long De Novo Lesions of Main Coronary Arteries (D-Lesion Long Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The People's Hospital of Liaoning Province (Other)
Responsible Party: Principal Investigator, Zhilin Miao, Vice-Director of Department of Cardiology, The People's Hospital of Liaoning Province
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTC-91919
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Stable Angina Pectoris; Unstable Angina Pectoris
Keywords: Drug-Coated Balloon; Main Coronary Artery; De Novo Lesion
MeSH Terms: conditions — Angina, Stable; Angina, Unstable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PCB group (Experimental): Prospective, single center, single-group clinical study. Interventions: Patients in the PCB group will be treated (angioplasted) with Paclitaxel-Coated Balloon (SeQuent ® Please; B.Braun, Melsungen, Germany)
  Interventions: Device: Paclitaxel-Coated Balloon

INTERVENTIONS:
Device: Paclitaxel-Coated Balloon — SeQuent ® Please; B.Braun, Melsungen, Germany
  Other Names: Drug-coated balloon (DCB)

SUMMARY:
This study evaluates the Efficacy and Safety of Paclitaxel-Coated Balloon Catheter in Patients With Diffuse Long De Novo Lesions of Main Coronary Arteries.

DETAILED DESCRIPTION:
Paclitaxel-Coated Balloon Catheter is a new device in coronary disease, it can inhibit the proliferation of smooth muscle of coronary vessels by transitory contaction, without residual implantation.

More and more evidences have shown its efficacy and safety in diffuse small coronary disease, bifurcation disease and in-stent restenosis. But there are still seldom evidences in De Novo Lesions of Main Coronary Arteries.

PCB has used in some subgroup of many study but confused with in-stent renstenosis or small coronary disease. The investigators designed this study to evaluate the Efficacy and Safety of Paclitaxel-Coated Balloon Catheter in Patients With Diffuse Long De Novo Lesions of Main Coronary Arteries.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of stable angina or unstable angina in hospitalized patients. Objective clinical evidence of ischemia (ECT, Exercise ECG, ECG ST-T changes) With CAG proven one vessel lesion（a lesion length of ≥ 20mm)；
2. a lesion diameter stenosis >75% as evaluated by QCA with a reference diameter of ≥ 2.75 mm and ≤ 3.5 mm .
3. a willingness or ability to provide informed consent，a willingness to receive telephone followed-up at postoperative 1 month, 3 month, 6 month, and an angiographic follow up at postoperative 9 month.
4. a willingness to receive DCB angioplast or DES implantation.

Exclusion Criteria:

1. Patients with acute myocardial infarction within 30 days；
2. a previous history of severe valvular heart disease,severe hepatic and renal insufficiency；severe cardiac dysfunction with EF≤40%；
3. advanced cancer with a life expectancy of <12 months；
4. Patients with abnormal coagulation function, Contraindications for antiplatelet drugs or unable to tolerate antiplatelet therapy;
5. Pregnant and lactating patients；
6. Multiple vessels involvement or multiple lesions requiring intervention treatment,left main artery lesions and coronary artery bypass graft lesions；
7. Stent restenosis
8. Thrombotic disease，severe calcified lesions（Judged by the operator， CAG showed class 2 or more severe calcified lesions），spontaneous dissection or ulcerative lesion，coronary ostial lesions (the lesion included should be an interval of greater than 3mm from the ostial of RCA or LAD)， severe angulated lesions（>45°）
9. diameter of collateral vessel≥ 2.25 mm requiring interventional therapy,type 1 coronary lesions（Patients with diameter of collateral vessel< 2.25 mm， who were not treated with DCB dilatation were also eligible）.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
QCA late lumen loss | Immediately after the procedure and at 9 months follow-up
  minimal lumen diameter at post-procedure minus minimal lumen diameter at 9 months follow-up measured by QCA(quantitative coronary angiography)

CONTACTS AND LOCATIONS:
Overall Officials: Aijie Hou, Principal Investigator — The People's Hospital of Liaoning Province
Locations (1):
- The People's Hospital of Liaoning Province, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided